CLINICAL TRIAL: NCT00636636
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Patients With Postherpetic Neuralgia
Brief Title: Safety and Efficacy of Gabapentin in Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81-0062; NCT01465321 (obsolete NCT alias)
Record Dates: First submitted 2008-02-21; First posted 2008-03-14 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Neuralgia,Postherpetic
Keywords: Postherpetic Neuralgia (PHN), shingles
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-ER (Experimental): Gabapentin - Extended Release
  Interventions: Drug: Gabapentin Extended Release tablets
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Extended Release tablets — Once-Daily; 300 mg and 600 mg tablets
  Arms: G-ER
Drug: Placebo — Once daily; 300 mg and 600 mg tablets
  Arms: Placebo

SUMMARY:
Gabapentin and pregabalin are treatments for some types of neuropathic pain, including postherpetic neuralgia (PHN). However, these treatments usually need to be taken 3 times a day for effective pain control. The purpose of this study is to determine whether a new gabapentin tablet, which only needs to be taken once a day, is safe and effective for the treatment of postherpetic neuralgia.

DETAILED DESCRIPTION:
The primary study objective is to assess the relative efficacy of G-ER dosed once daily (1800 mg following the evening meal), versus placebo in reducing the mean daily pain score from the baseline week to the end of the efficacy treatment period (Treatment Week 10) in patients with PHN.

Secondary efficacy measures will include changes from baseline in mean weekly sleep interference scores, Short-Form McGill Pain Questionnaire (SF-MPQ), the Neuropathic Pain Scale (NPS), Brief Pain Inventory (BPI), Patient Global Impression of Change (PGIC), and Investigator-Rated Clinical Global Impression of Change (CGIC).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years or older who have experienced pain for at least 6 months, but not more than 5 years after the healing of a herpes zoster skin rash(typically about 4 months after the rash first appears).
2. Patient has a pain intensity score of at least 4 on the 11-point Numerical Rating Scale (NRS). Patients should never be informed of the pain intensity criterion prior to screening or randomization.
3. Patients of child-bearing potential must have a negative serum pregnancy test at screening and a negative follow-up urine pregnancy test at randomization.
4. Patient has a mean baseline week pain intensity score of at least 4 on the 11-point NRS scale at the end of a 1-week baseline period and has completed at least 4 days of daily pain diary entries during the baseline week.
5. Patients must have a minimum washout period of greater than 5 times the half-life of the drug of several medications.
6. Patients currently treated with gabapentin pr pregabalin at screening may be eligible for the study, but must have a tapering period wherein the dose of gabapentin or pregabalin is reduced gradually over a period of 5 days followed by a two day washout prior to the Baseline Week.

Exclusion Criteria:

1. Patients who have previously not responded to treatment for PHN with gabapentin or pregabalin.
2. Patients who previously experienced dose-limiting adverse effects that prevented titration of gabapentin to an effective dose.
3. Patient is a nursing mother.
4. Patient has hypersensitivity to gabapentin.
5. Patient has had neurolytic or neurosurgical treatment for PHN.
6. Patient has severe pain from causes other than PHN.
7. Patient has used injected anesthetics or steroids within 30 days of baseline.
8. Patient has skin conditions in the area affected by the neuropathy that could alter sensation.
9. Patient is in an immunocompromised state.
10. Patient has an estimated creatinine clearance less than 50 ml/min.
11. Patient has had malignancy within past 2 years other than basal cell carcinoma.
12. Patient has had gastric reduction surgery.
13. Patient has severe chronic diarrhea, chronic constipation [unless attributed to drugs that will be washed out], uncontrolled irritable bowel syndrome (IBS) or unexplained weight loss.
14. Patient has any abnormal chemistry or hematology results that are deemed by the investigator to be clinically significant.
15. Patient has a history of substance abuse within the past year.
16. Patient has a history of seizure (except for infantile febrile seizure) or is at risk of seizure due to head trauma.
17. Patient has a history of chronic hepatitis B or C, hepatitis within the past 3 months, or HIV infection.
18. Patient has any other clinically significant medical or psychological condition that, in the opinion of the Investigator would jeopardize the safety of the patient or affect the validity of the study results.
19. Continuing use of any concomitant medication excluded by Inclusion Criterion 5.
20. Patient has participated in a clinical trial of an investigational drug or device within 30 days of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (36):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Lancaster, California
  - Los Angeles, California
  - Pismo Beach, California
  - Colorado Springs, Colorado
  - Pueblo, Colorado
  - Daytona Beach, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Elk Grove Village, Illinois
  - Shreveport, Louisiana
  - West Yarmouth, Massachusetts
  - Ann Arbor, Michigan
  - Florissant, Missouri
  - Jefferson City, Missouri
  - Albuquerque, New Mexico
  - High Point, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Kettering, Ohio
  - Warwick, Rhode Island
  - Murrells Inlet, South Carolina
  - Pelzer, South Carolina
  - Tullahoma, Tennessee
  - Austin, Texas
  - Longview, Texas
  - Spokane, Washington
- Buenos Aires, Argentina
- Russia (2):
  - All Over Russia
  - Saint Petersburg

REFERENCES:
- [Derived] Mehta N, Bucior I, Bujanover S, Shah R, Gulati A. Relationship between pain relief, reduction in pain-associated sleep interference, and overall impression of improvement in patients with postherpetic neuralgia treated with extended-release gabapentin. Health Qual Life Outcomes. 2016 Apr 1;14:54. doi: 10.1186/s12955-016-0456-0. PMID 27037091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from March 2008 through May 2009.
Pre-assignment Details: Study included screening visit, wash-out from all PHN medications as necessary, followed by a week of baseline period. Patients who successfully completed the baseline week, if still continues to meet entry criteria, then get randomized to Active or Placebo groups.
Groups:
- G-ER: Gabapentin Extended Release 1800 mg once daily (qd); 300 mg and 600 mg tablets, oral dosing
- Placebo: Placebo 1800 mg once daily (qd); 300 mg and 600 mg sugar pills, oral dosing
Period: Overall Study
Arm/Group | G-ER | Placebo
Started | 221 | 231
Safety & Efficacy of Gabapentin ER | 186 | 194 (1 patient randomized twice, not included in ITT, but completed medication and counted as completer)
379 | 186 | 194 (1 patient randomized twice, not included in ITT, but completed medication and counted as completer)
Completed | 185 | 192
Not Completed | 36 | 39
Not completed — Other reason | 4 | 6
Not completed — Adverse Event | 19 | 8
Not completed — Lack of Efficacy | 7 | 12
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-ER | Placebo | Total
Number analyzed (Participants) | 220 | 230 | 450
Age Continuous [Mean (Standard Deviation); unit: years] | 65.3 (13.3) | 65.9 (11.1) | 65.6 (12.2)
Age, Customized [Number; unit: participants] — Of the 452 subjects randomized, 2 subjects were excluded from the intent-to-treat (ITT) population: 1 subject had no baseline data recorded, and 1 subject was randomized twice. Baseline demographics were calculated on the ITT population of 450 participants.
  participants
    <65 years | 81 | 89 | 170
    65 to 74 years | 82 | 86 | 168
    >=75 years | 57 | 55 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 147 | 281
  Male | 86 | 83 | 169
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 196 | 204 | 400
  Black | 10 | 6 | 16
  Asian | 1 | 2 | 3
  Other | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Baseline Observation Carried Forward (BOCF) Average Daily Pain Score
Description: Average daily pain scored on 11-point numerical rating scale (where 0 = no pain, 10 = worst possible pain). Results presented as least squares (LS) mean change in baseline observation carried forward (BOCF) average daily pain score from baseline to the final week of efficacy treatment period (Week 10).
Time Frame: 10 weeks
Population: ITT, BOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | G-ER | Placebo
Number analyzed (Participants) | 220 | 230
Scores on a scale | -2.12 (0.17) [-2.44 to -1.79] | -1.63 (0.16) [-1.95 to -1.30]
Statistical Analysis 1: Comparison: G-ER vs Placebo; Test type: Superiority or Other; p = 0.0125, ANCOVA; Least squares mean difference = -0.49, 95% CI 2-sided [-0.88 to -0.11], Standard Error of Mean 0.20

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient self-assessment of how much pain had changed at end of treatment period (Week 10) compared to pain at baseline; scored on 7-point numerical rating scale (where 1 = very much improved, 7 = very much worse). Results presented as number of participants categorized at end of treatment (Week 10) as "very much improved" (score = 1) or "much improved" (score = 2).
Time Frame: 10 weeks
Population: ITT, BOCF
Measure: Number; unit: Participants
Arm/Group | G-ER | Placebo
Number analyzed (Participants) | 220 | 230
Participants | 94 | 77
Statistical Analysis 1: Comparison: G-ER vs Placebo; P-value (vs Placebo) for pairwise test of treatment effect between G-ER group and Placebo group is based on Z test for difference between the 2 groups in proportion of participants who were categorized as very much or much improved in PGIC at endpoint. Proportion in each group calculated from number of participants categorized as very much or much improved relative to total number of participants in ITT population; Test type: Superiority or Other; p = 0.0434, Z test; Difference in proportion = 0.092, 95% CI 2-sided [-0.00 to 0.18]

3. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: Investigator assessment of patient's overall PHN symptoms at end of treatment period (Week 10) compared to overall PHN symptoms at baseline; scored on 7-point numerical rating scale (where 1 = very much improved, 7 = very much worse). Results presented as number of participants categorized at end of treatment (Week 10) as "very much improved" (score = 1) or "much improved" (score = 2).
Time Frame: 10 weeks
Measure: Number; unit: Participants
Arm/Group | G-ER | Placebo
Number analyzed (Participants) | 220 | 230
Participants | 97 | 78
Statistical Analysis 1: Comparison: G-ER vs Placebo; P-value (vs Placebo) for pairwise test of treatment effect between G-ER group and Placebo group is based on Z test for difference between the 2 groups in proportion of participants who were categorized as very much or much improved in CGIC at endpoint. Proportion in each group calculated from number of participants categorized as very much or much improved relative to total number of participants in ITT population; Test type: Superiority or Other; p = 0.0268, Z test; Difference in proportion = 0.102, 95% CI 2-sided [0.01 to 0.19]

4. Secondary Outcome: Average Daily Sleep Interference Score
Description: Assessed on 11-point numeric rating scale (where 0 = pain does not interfere with sleep, 10 = pain completely interferes with sleep); evaluated from daily sleep entry in electronic diary. Results presented as least squares (LS) mean change in baseline observation carried forward (BOCF) average daily sleep interference score from baseline to final week of treatment period (Week 10).
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | G-ER | Placebo
Number analyzed (Participants) | 220 | 230
Scores on a scale | -2.30 (0.16) | -1.59 (0.15)
Statistical Analysis 1: Comparison: G-ER vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Least square mean difference = -0.71, 95% CI 2-sided [-1.07 to -0.35], Standard Error of Mean 0.18 — P-value versus Placebo for pairwise test of difference of LS mean change from baseline between G-ER and Placebo groups is based on t-test of Type III analysis

5. Other Pre Specified Outcome: Mean Change in Last Observation Carried Forward (LOCF) Average Daily Pain Score
Description: Average daily pain scored on 11-point numerical rating scale (where 0 = no pain, 10 = worst possible pain). Results presented as least squares (LS) mean change in last observation carried forward (LOCF) average daily pain score from baseline to final week of efficacy treatment period (Week 10).
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | G-ER | Placebo
Number analyzed (Participants) | 220 | 230
Scores on a scale | -2.40 (0.17) | -1.85 (0.17)
Statistical Analysis 1: Comparison: G-ER vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Least square mean difference = -0.55, 95% CI 2-sided [-0.96 to -0.15], Standard Error of Mean 0.20

ADVERSE EVENTS:
Time Frame: 11 weeks (plus 30 days for SAEs)
Description: AEs and SAEs collected from signing of consent form through completion of Tapering Week Visit (Week 11); SAEs collected for 30 days after completion of Tapering Week (Week 11).
Arm/Group | G-ER | Placebo
Serious Adverse Events (participants affected / at risk) | 4/221 | 6/231
Other Adverse Events (participants affected / at risk) | 92/221 | 63/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER (N=221) | Placebo (N=231)
Cardiac failure congestion (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Left arm fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancoast tumor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER (N=221) | Placebo (N=231)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Blood pressure increased (Investigations) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 5 (5)
Dizziness (Nervous system disorders) | 25 (25) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 10 (10) | 9 (9)
Herpes zoster (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 10 (10) | 7 (7)
Peripheral edema (General disorders) | 7 (7) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 2 (2) | 4 (4)
Somnolence (Nervous system disorders) | 12 (12) | 7 (7)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Weight increased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agree that the sponsor shall have the right to the first publication of the results of the study which is intended to be joint, multi-center publication. Following the first publication, the PI may publish data or results from the study, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the data of the proposed publication.Sponsor may remove any information that is considered confidential and or proprietary other than study data.